CLINICAL TRIAL: NCT05295615
Title: Effects of PEMF Treatment on Patients With Mild to Moderate Alzheimer's Disease in a Controlled Pilot Study
Brief Title: Pulsed Electromagnetic Field Treatment In Patients With Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herrick Medical LLC (Industry)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM003
Record Dates: First submitted 2022-02-15; First posted 2022-03-25 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active ECHS AD device (Experimental): Experimental intervention arm
  Interventions: Device: ECHS AD Device

INTERVENTIONS:
Device: ECHS AD Device — Pulsed electromagnetic therapy device

SUMMARY:
An open label pilot study in mild to moderate AD patients to assess the effects of treatment with ECHS AD pulsed electromagnetic treatment device on disease progression. Enrolled patients will receive active devices. They will treat themselves at home three times a day for 15 minutes over 120 days. Primary end points are the The Alzheimer's Disease Assessment Scale-Cognitive Subscale and the Mini-Mental State Exam. Participants will be followed-up for 9 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years
2. Patients diagnosed with mild to moderate Alzheimer's Dementia defi
3. At least an eighth grade of educational achievement
4. If female, post-menopausal.
5. MMSE score between 16 and 26
6. Capable of providing consent or having a surrogate (e.g., spouse, family member) capable of providing consent if participant lacks consent capacity
7. Able and willing to comply with the protocol
8. If the participant is receiving a cholinesterase inhibitor and/or memantine, such medication has been prescribed for at least 3 months prior to screening and the dose is stable for at least 60 days prior to screening (that dose needs to be maintained throughout the period of this study)
9. Spouse, family member or professional caregiver agree and are capable of taking care of the participation of the patient in the study (answering questions regarding the patient's condition, assuming responsibility for medication, and applying and supervising the daily PEMF treatments)
10. Physical clearance for study participation as evaluated by the clinician

Exclusion Criteria:

1. The patient lacks capacity to consent to study participation and no surrogate is available to provide consent
2. History of epileptic seizures or epilepsy
3. Currently taking medication that lowers the seizure threshold
4. Presence of depression, bipolar disorder, a psychotic disorder, or any other neurological or psychiatric condition (whether now or in the past), which the Investigator finds as interfering with the study
5. Severe agitation that would interfere with study procedures
6. Alcoholism or substance use disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
7. Major surgery (defined as any major abdominal, vascular or thoracic surgery requiring general anesthesia and resulting in a period of >1 week hospitalization) within 4 weeks
8. Head anatomy that interferes with the fit of the treatment device
9. Participation in another clinical trial within the previous 30 days
10. Metal implants in the head, (i.e., cochlear implants, implanted brain stimulators and neurostimulators, aneurysm clips) with the exception of metal implants in mouth

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | Change between day 0, and 30, 60, 90, 120, 150, 240, 310, 400 days
  Assessment consisting of 11 tasks, taking up to 30mins, to measure the severity of cognitive dementia symptoms. Score 0-70, Higher number, more severity.
Mini-Mental Status Exam (MMSE) | Change between day 0, and 30, 60, 90, 120, 150, 240, 310, 400 days
  Clinician assessment of cognitive impairment. Scoring 0-30, lower score, more severity
Global Deterioration questionnaire | Change between day 0, and 30, 60, 90, 120, 150, 240, 310, 400 days
  Clinician assessment of cognitive impairment. Scored 0-7, higher score, greater severity
Quality of Life Scale | Change between day 0, and 30, 60, 90, 120, 150, 240, 310, 400 days
  Clinician assessment of cognitive impairment. Scored 0-7, higher score, greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- Hackensack Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided